CLINICAL TRIAL: NCT07198373
Title: Exploratory Study on the Efficacy of Zebutinib as Maintenance Therapy Following CAR-T Cell Therapy in Patients With Non-Hodgkin B-Cell Lymphoma
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Kai Hu, Director of the Lymphoma Department at Beijing Gao Bo Hospital, Beijing GoBroad Hospital
Other Study IDs: GBYY2527
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance Therapy Group
  Interventions: Drug: Maintenance Therapy Group

INTERVENTIONS:
Drug: Maintenance Therapy Group — Patients achieving remission (complete or partial) at the 3-month post-CAR-T infusion assessment receive oral zanubrutinib capsules for maintenance therapy for 2 years.

SUMMARY:
This study is a single-center, Phase IV clinical trial designed to collect and analyze data on the efficacy and safety of zanubrutinib as maintenance therapy following CAR-T cell therapy in subjects with non-Hodgkin B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years, no gender restrictions; (2) Expected survival time exceeding 12 weeks; (3) Cytologically or histopathologically confirmed diagnosis of non-Hodgkin B-cell lymphoma according to WHO 2016 criteria; (4) Platelet count ≥ 50 × 10⁹/L; (5) Currently undergoing or scheduled to initiate oral zanubrutinib maintenance therapy following autologous or allogeneic CAR-T cell therapy; (6) Able to understand this trial and has signed an informed consent form.

Exclusion Criteria:

* (1) Pregnant or lactating individuals; male subjects planning to conceive within one year of treatment or within one year after cell reinfusion, or whose partners plan to conceive within one year after cell reinfusion; (2) Individuals with medical conditions that affect their ability to sign a written informed consent form or comply with study procedures; or those unwilling or unable to adhere to study requirements; (3) Individuals deemed unsuitable for participation in this trial by the investigator.

  1. Pregnant or lactating individuals; or male subjects planning to conceive within one year of treatment or within one year after cell infusion, or whose partners plan to conceive within one year after cell infusion; (2) Individuals with medical conditions that prevent signing a written informed consent form or complying with study procedures; or those unwilling or unable to comply with study requirements; (3) Individuals deemed unsuitable for this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who achieve remission (complete or partial) at the 3-month post-CAR-T infusion assessment
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 24 months post-administration | From date ofrandomization untilhe date of first documented progression , assessed up to 24 months

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | The time from the start of cell infusion to the first assessment of progression or death from any cause， assessed up to 5 years
Overall Survival (OS) | From date of randomization untilhe date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years

IPD SHARING:
Plan to Share IPD: No